CLINICAL TRIAL: NCT00213512
Title: Traitment of Patients Presenting Pemphigus With Anti CD20 (Mabthera).
Brief Title: Effect of Anti CD20 in Pemphigus Desease
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2002/020/HP
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2013-06-18 (Estimated); Status verified 2013-06

CONDITIONS: Pemphigus
MeSH Terms: conditions — Pemphigus | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Mabthera

SUMMARY:
to treat in an open non comparative clinical study patients presenting pemphigus with corticodependance, corticoresistance and contre-indication to systemic steroids.

ELIGIBILITY:
Inclusion Criteria:

* age>18
* pemphigus corticoresistant
* pemphigus cortico dependant
* contre-indications : systémic steroids

Exclusion Criteria:

* age < 18
* cardiopathie
* pregnant woman
* absence contraception
* no consentment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22
Dates: Start 2003-06; Primary Completion 2006-06 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
primary end-point was the rate of CR three months after the last infusion of Rituximab

SECONDARY OUTCOMES:
secondary end-points were :
rate of CR during the study period
time from the start of Rituximab to CR
number and length of time to relapses
treatment tolerance

CONTACTS AND LOCATIONS:
Overall Officials: pascal Joly, MD-PHD, Principal Investigator — UH-Rouen
Locations (1):
- UH-Rouen, Rouen, Seine maritime, France

REFERENCES:
- [Derived] Joly P, Mouquet H, Roujeau JC, D'Incan M, Gilbert D, Jacquot S, Gougeon ML, Bedane C, Muller R, Dreno B, Doutre MS, Delaporte E, Pauwels C, Franck N, Caux F, Picard C, Tancrede-Bohin E, Bernard P, Tron F, Hertl M, Musette P. A single cycle of rituximab for the treatment of severe pemphigus. N Engl J Med. 2007 Aug 9;357(6):545-52. doi: 10.1056/NEJMoa067752. PMID 17687130